CLINICAL TRIAL: NCT05107245
Title: Observational Study on the Diagnostic Evaluation of the Intestinal Microbiota of French People Infected With the SARS-CoV-2.
Brief Title: Observational Study on the Diagnostic Evaluation of the Intestinal Microbiota of Patients With COVID-19.
Acronym: EDIFICE
Status: Completed | Type: Observational
Sponsor: Luxia Scientific (Industry)
Collaborators: Clinique Saint Jean Ermitage (Unknown); Nantes University Hospital (Other); Centre Hospitalier de Fontainebleau (Unknown); Clinique du Mousseau (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2020-A00979-30
Record Dates: First submitted 2021-10-22; First posted 2021-11-04 (Actual); Last update posted 2021-12-20 (Actual); Status verified 2021-12

CONDITIONS: COVID-19
Keywords: microbiome ; SARS-CoV-2 ; metagenomic ; stool
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stool
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COVID-19 patients: Hospitalised COVID-19 patients
  Interventions: Diagnostic Test: 1test1
- Controls: Exposed medical staff
  Interventions: Diagnostic Test: 1test1

INTERVENTIONS:
Diagnostic Test: 1test1 — Loss of bacterial diversity diagnosis

SUMMARY:
In the context of the COVID-19 pandemic, the role of the gut microbiome is yet unknown. The aim of this trial is to evaluate the clinical contribution of the gut microbiome composition and diversity on the disease severity and to estimate the viral load in stool samples.

ELIGIBILITY:
Inclusion Criteria:

* COVID-19 positive patients: hospitalised patients diagnosed with COVID-19 in one of the investigating sites, and able to provide a stool sample.
* Control subjects: Medical and paramedical personnel working at one of the investigating sites, having been in direct contact with the patients.
* Aged between 18 and 95 years.
* Subjects able to read the French-language study information leaflet.
* Patients with social cover.

Exclusion Criteria:

* COVID-19 negative patients.
* Patients in critical care, heart failure or respiratory failure.
* Unable to provide naturally a stool sample.
* Patients without social cover.
* Pregnant women

Ages: 18 Years to 95 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: COVID-19 positive patients: hospitalised patients diagnosed with COVID-19 in one of the investigating sites, and able to provide a stool sample.
  + Control subjects: Medical and paramedical personnel working at one of the investigating sites, having been in direct contact with the patients.
Sampling Method: Non-Probability Sample
Enrollment: 143 (Actual)
Dates: Start 2020-04-28 (Actual); Primary Completion 2021-04-29 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Alpha-diversity | at the time of inclusion in the study
  Alpha-diversity of the gut microbiota measured by 16S sequencing

SECONDARY OUTCOMES:
SARS-CoV-2 load | at the time of inclusion in the study
  SARS-CoV-2 load in stool measured by RT-PCR
Microbiome composition | at the time of inclusion in the study
  Genus level of the gut microbiota measured by 16S sequencing

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - Centre Hospitalier Universitaire de Nantes, Nantes, Pays de la Loire Region
  - Centre Hospitalier de Fontainebleau, Fontainebleau, Seine-et-Marne
  - Clinique Saint Jean l'Ermitage, Melun, Seine-et-marne
  - Clinique du Mousseau, Évry-Courcouronnes, Île-de-France Region

IPD SHARING:
Plan to Share IPD: Yes